CLINICAL TRIAL: NCT01259557
Title: Multi-center, Phase Ⅳ, Single Arm, Open-label Clinical Trial to Evaluate the Efficacy and Safety of Meditoxin® in Subjects With Essential Blepharospasm
Brief Title: Efficacy and Safety Study of Meditoxin® to Treat Essential Blepharospasm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Yujin Sun / CRA, Medytox
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-PRT-BP02
Record Dates: First submitted 2010-11-25; First posted 2010-12-14 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Essential Blepharospasm
MeSH Terms: conditions — Benign essential blepharospasm | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum toxin type A(Meditoxin®) (Experimental)
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 2 times, Intra-muscular injection, Maximum dosage total 60U
  Other Names: Meditoxin; Neuronox

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Meditoxin® in the treatment of Essential blepharospasm.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged above 18
* Subjects who was diagnosed with Essential Blepharospasm
* Subjects who voluntarily Signed written informed consent
* Subjects who can adhere to protocol and study requirements

Exclusion Criteria:

* Subjects with known history of allergy considered due to Botulinum toxin type A
* Subjects who have received botulinum toxin A type within 3 months
* Any disease that might affect neuromuscular function (e.g.. Myasthenia Gravis, Lambert-Eaton Syndrome, Amyotrophic Lateral Sclerosis ect.)
* Subjects who are participating in other clinical trials
* Pregnant or lactating female Subjects
* Subjects who are not eligible for the study at the discretion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
the change rate of Jankovic Rating Scale score | 4weeks
  To evaluate the change of JRS(Jankovic Rating Scale) score at 4 weeks post treatment based on baseline( 0 week).

SECONDARY OUTCOMES:
the change rate of Jankovic Rating Scale scale | 0 week, 16weeks(or retreatment point)
  To evaluate the change of JRS(Jankovic Rating Scale) at retreatment point or 16 weeks post treatment based on Baseline(0 week).
the change rate of Blepharospasm Disability Index | 0week, 4weeks, 8weeks, 16weeks(or retreatment point)
  To evaluate the change of Blepharospasm Disalbility Index at 4weeks, 8weeks, 16weeks(or retreatment point) post treatment.
Global assessment about the improvement | 4weeks
  To evaluate the Global assessment about the improvement at 4weeks post treatment.
the duration of efficacy | retreatment point or 16 weeks
  To evaluate the duration of efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jaechan Kim, M.D., Ph.D., Principal Investigator — Chung-Ang university Yongsan Hospital
Locations (3):
- South Korea (3):
  - Sevrance Hospital, Seoul
  - Seoul St.Mary Hospital, Seoul
  - Chung-Ang Univesity Yongsan Hospital, Seoul